CLINICAL TRIAL: NCT01071109
Title: The Clinical and Biochemical Effect of Therapeutic Massage on Fatigue and Insomnia in Women With Breast Cancer Receiving Radiation Therapy
Acronym: RTTM301
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Floyd Memorial Hospital and Health Services (Other)
Collaborators: Indiana University (Other)
Responsible Party: Judith G. Myers, PhD, Indiana University Southeast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTTM301
Record Dates: First submitted 2010-02-16; First posted 2010-02-19 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer; Fatigue; Insomnia
Keywords: Therapeutic massage; massage; inflammation; fatigue; insomnia; radiation therapy; breast cancer; Breast Cancer patients receiving radiation therapy
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Sleep Initiation and Maintenance Disorders; Inflammation | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Massage (Experimental)
  Interventions: Procedure: Therapeutic Massage
- No therapeutic massage (No Intervention)

INTERVENTIONS:
Procedure: Therapeutic Massage — Therapeutic Massage--subjects randomized to this group will receive weekly, one-hour therapeutic massage
  Arms: Therapeutic Massage

SUMMARY:
A majority of women with breast cancer receive radiation therapy, and many of them experience the debilitating side effects of fatigue and insomnia. There is a need for an effective treatment that could ameliorate these symptoms and improve quality of life in the radiation therapy population.

The primary purpose of the proposed research is to study the impact of massage therapy as a tool for the management of fatigue and insomnia experienced by women diagnosed with breast cancer and receiving radiation therapy.

The secondary purpose is to explain, at the biochemical level, the effect of therapeutic massage on the level of fatigue and insomnia in radiation therapy patients. Prior studies have shown an association between fatigue and insomnia in the breast cancer patient following radiation therapy and the presence of inflammation as evidenced by increased proinflammatory cytokine production. The investigators hypothesize that therapeutic massage will ameliorate the symptoms of fatigue and insomnia associated with radiation therapy, and will be associated with a reduction in the plasma levels of interleukin-6 (IL-6),soluble IL-6 receptor (sIL-6R/CD126), and C-Reactive Protein (CRP). This reduction in proinflammatory biomarkers will be due to the activation of the cholinergic anti-inflammatory pathway via the activation of the vagus nerve.

ELIGIBILITY:
Inclusion Criteria:

* female patients and
* > or = 18 years of age and
* diagnosed with breast cancer and
* undergoing radiation therapy and
* willing to follow protocol requirements

Exclusion Criteria:

* Stage IV disease or
* Presence of an underlying disease that is anticipated to be fatal w/in 6 mo
* Long term steroid medications in the past year or
* Plans to move out of study region within six months or
* Receiving regular body work over the past six months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-10 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Fatigue Symptom Inventory, Pittsburgh Sleep Quality Index, and Insomnia Severity Index scores over time. | Baseline, End of Treatment (6 weeks), End of Study (3 months after End of Treatment)

SECONDARY OUTCOMES:
Plasma levels of proinflammatory markers: interleukin-6 (IL-6), soluble IL-6 receptor (sIL-6R/CD126), and C-Reactive Protein (CRP). | Baseline, End of Treatment (6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G Myers, PhD, Principal Investigator — Indiana University Southeast
Locations (1):
- FMHHS Cancer Care Center, New Albany, Indiana, United States